CLINICAL TRIAL: NCT00995215
Title: Evaluation of Wire Electrodes to Activate the Expiratory Muscles to Restore Cough
Brief Title: Sub-study to Spinal Cord Stimulation to Restore Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Anthony F. Dimarco, Professor of Medicine, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB08-00269/IRB98-00091; IRB08-00269 (Other: IRB); IRB98-00091 (Other: IRB)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough
Keywords: spinal cord injury; paralysis; cough; cervical spinal cord injury; thoracic spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal Cord Stimulation (Experimental): The participant will have wire electrodes temporarily placed - by a routine surgical procedure - over the surface of the spinal cord on the lower back. These electrodes will be activated in the operating room and the degree of muscle activation assessed. The wire electrodes will then be removed. Small, disc electrodes will then be permanently implanted to stimulate expiratory muscles and restore cough. These electrodes are activated using an external control unit.
  Interventions: Procedure: Spinal Cord Stimulation; Device: Expiratory Muscle Stimulator

INTERVENTIONS:
Procedure: Spinal Cord Stimulation — The participant will have wire electrodes temporarily placed - by a routine surgical procedure - over the surface of the spinal cord on the lower back. These electrodes will be activated in the operating room and the degree of muscle activation assessed. The wire electrodes will then be removed. Small, disc electrodes will then be permanently implanted to stimulate expiratory muscles and restore cough. These electrodes are activated using an external control unit.
  Other Names: NeuroControl Expiratory Muscle Stimulation (IDE G980267)
Device: Expiratory Muscle Stimulator — The expiratory muscle stimulator consists of three small electrodes (metal discs) implanted over the surface of their spinal cords on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.

SUMMARY:
Evaluation of Wire Electrodes to Activate the Expiratory Muscles to Restore Cough

DETAILED DESCRIPTION:
Patients with cervical and thoracic spinal cord injuries often have paralysis of a major portion of their expiratory muscles - the muscles responsible for coughing - and therefore, lack a normal cough mechanism. Consequently, most of these patients suffer from a markedly reduced ability to clear airway secretions, a factor which contributes to the development of recurrent respiratory tract infections such as pneumonia and bronchitis. In fact, pneumonia is a major cause of death in this patient population.

In a recent clinical trial, we have shown that the expiratory muscles can be electrically activated by spinal cord stimulation (SCS), a technique which involves the surgical placement of disc electrodes on the surface of the spinal cord. This method is successful in achieving an effective means of expiratory muscle activation, as demonstrated by the generation of large airway pressures and peak airflow rates. Importantly, SCS facilitates secretion removal, reduces the need for caregiver support, reduces the incidence of respiratory tract infections and improves life quality. This method therefore has the potential to reduce health care costs and improve survival in spinal cord injured subjects.

The purpose of this trial is to directly compare activation of the expiratory muscles using wire electrodes, which can be inserted percutaneously through a needle, with the previously employed disc electrodes.

In this trial, researchers will study 6 adults (18-70 years old) with spinal injuries (T5 level or higher), at least 12 months following the date of injury. After an evaluation including medical history, a brief physical examination, and initial testing, each participant will undergo a surgical procedure to implant small electrodes (metal discs) over the surface of the spinal cord on the lower back to stimulate the expiratory muscles and restore cough. Prior to permanent implantation of this system, wire and disc electrodes will be compared by assessing the degree of expiratory muscle activation with each electrode type. The disc electrodes will then be permanently implanted, allowing the participant to have use of a fully functioning stimulation system to restore an effective cough.

ELIGIBILITY:
Inclusion Criteria:

* Stable spinal cord injury T5 level or higher
* Expiratory muscle weakness

Exclusion Criteria:

* Significant cardiovascular disease
* Active lung disease
* Brain disease
* Scoliosis, chest wall deformity, or marked obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10; Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F. DiMarco, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Spinal cord stimulation: a new method to produce an effective cough in patients with spinal cord injury. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1386-9. doi: 10.1164/rccm.200601-097CR. Epub 2006 Mar 16. PMID 16543552
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-sponsored clinical trial. Part I: methodology and effectiveness of expiratory muscle activation. Arch Phys Med Rehabil. 2009 May;90(5):717-25. doi: 10.1016/j.apmr.2008.11.013. PMID 19406289
- [Result] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR, Frost FS, Creasey GH, Nemunaitis GA. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-Sponsored clinical trial. Part II: clinical outcomes. Arch Phys Med Rehabil. 2009 May;90(5):726-32. doi: 10.1016/j.apmr.2008.11.014. PMID 19406290

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation: The participant will have wire electrodes temporarily placed - by a routine surgical procedure - over the surface of the spinal cord on the lower back. These electrodes will be activated in the operating room and the degree of muscle activation assessed. The wire electrodes will then be removed. Small, disc electrodes will then be permanently implanted to stimulate expiratory muscles and restore cough. These electrodes are activated using an external control unit
  Spinal Cord Stimulation: The participant will have wire electrodes temporarily placed - by a routine surgical procedure - over the surface of the spinal cord on the lower back. These electrodes will be activated in the operating room and the degree of muscle activation assessed. The wire electrodes will then be removed. Small, disc electrodes will then be permanently implanted to stimulate expiratory muscles and restore cough. These electrodes are activated using an external control unit.
  Expiratory Muscle Stimulator: T
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: These studies were performed in subjects (n=6) undergoing surgery for permanent placement of disc electrodes to restore cough in our previous clinical trial.
Groups:
- Evaluation of Temporary, Intra-operative Wire Lead Placement i: These studies were performed in subjects (n=6) undergoing surgery for permanent placement of disc electrodes to restore cough in our previous clinical trial
Arm/Group | Evaluation of Temporary, Intra-operative Wire Lead Placement i
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.6 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Patient with cervical spinal cord injury [Count of Participants; unit: Participants] — The purpose of this study is to evaluate the efficacy of a wire electrode design temporarily placed during the surgical procedures for study 98-00091. The wire electrodes and the disc electrodes [currently in use] are each tested intra-operatively, and the results compared
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: The Effects of Electrical Spinal Cord Stimulation (SCS) on Airway Pressure Generation While Using Temporarily Placed Parallel Wire Leads and Implanted Disc Electrodes
Description: The effects of SCS with temporarily placed parallel wire leads and then with permanently implanted disc electrodes on airway pressure generation in each participant was evaluated in the operating room. The wire electrodes were temporarily placed (immediately prior to placement of disc electrodes as part of the current clinical trial) over the surface of the spinal cord on the lower back. These electrodes were activated, and the degree of expiratory muscle activation were assessed. The wire electrodes were then removed. Small, disc electrodes were then permanently implanted to stimulate expiratory muscles and restore cough. All measurements were repeated. Since SCS with the disc electrode leads, when applied in clinical trials, resulted in airway pressure generation that approximated pressures generated with a normal maximum cough, airway pressure generation achieved during SCS with these leads served as our gold standard to which all comparisons were made.
Time Frame: intra-operative
Population: Patients with spinal cord injury with expiratory muscle paralysis.
Measure: Mean (Standard Error); unit: cmH2O
Groups:
- Spinal Cord Stimulation (SCS) With Disc Electrodes: Effects of electrical spinal cord stimulation with disc on airway pressure generation was evaluated.
- Spinal Cord Stimulation (SCS) With Parallel Wire Leads: Effects of electrical spinal cord stimulation (SCS) with parallel wire leads on airway pressure generation was evaluated.
Arm/Group | Spinal Cord Stimulation (SCS) With Disc Electrodes | Spinal Cord Stimulation (SCS) With Parallel Wire Leads
Number analyzed (Participants) | 6 | 6
cmH2O | 56 (13) | 54 (9)
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) With Disc Electrodes vs Spinal Cord Stimulation (SCS) With Parallel Wire Leads; The effects of electrical (spinal cord stimulation) SCS with disc electrode and wire leads on airway pressure generation were compared. Since SCS with the disc leads, when applied in clinical trials, resulted in airway pressure generation that approximated pressures generated with a normal maximum cough, airway pressure generation achieved during SCS with these leads served as our gold standard to which all comparisons were made; Test type: Other — Statistical analysis was performed using a repeated measures analysis of variance and paired t-test; p = 0.05, ANOVA — A P value <0.05 was taken as indicative of statistical significance

ADVERSE EVENTS:
Time Frame: intra-operative
Description: No Adverse Events reported
Groups:
- Spinal Cord Stimulation: Experimental: Spinal Cord Stimulation
  The participant will have wire electrodes temporarily placed - by a routine surgical procedure - over the surface of the spinal cord on the lower back. These electrodes will be activated in the operating room and the degree of muscle activation assessed. The wire electrodes will then be removed. Small, disc electrodes will then be permanently implanted to stimulate expiratory muscles and restore cough. These electrodes are activated using an external control unit.
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2011-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT00995215/SAP_000.pdf
  • Informed Consent Form (2008-07-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT00995215/ICF_001.pdf
  • Study Protocol (2008-07-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT00995215/Prot_002.pdf